CLINICAL TRIAL: NCT02884349
Title: An Investigation of the Relationship Between Total Hip Implant Position and Hip Range of Movement
Brief Title: The Relationship Between Component Position and RoM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Ortho 15-08
Record Dates: First submitted 2016-05-18; First posted 2016-08-31 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Arthropathy of Hip
Keywords: Computer aided orthopaedic surgery; Implant orientation; Range of motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RoM assessment (Experimental): All patients recruited to the study.
  Interventions: Procedure: RoM assessment

INTERVENTIONS:
Procedure: RoM assessment — This group will have a CT scan at three months post-operatively instead of the two radiographs, an anterior/posterior pelvis view and a lateral hip view, which are standard care. They will also have a RoM assessment session in the movement analysis laboratory in the hospital at the same time point lasting about one hour, which is additional to standard care.

SUMMARY:
The aim of the study is to determine the influence of the combined anteversion of acetabular cup and the femoral stem used in total hip arthroplasty on the theoretical and actual range of motion of the hip in three dimensional space.

DETAILED DESCRIPTION:
Ninety patients from the clinics of a single consultant orthopaedic surgeon, who are listed to for total hip arthroplasty will be recruited to the study. They will have their surgery performed by the participating consultant as per his standard practice for the target study patient. This involves using the Excia T cementless stem, the ceramic femoral head, the Plasmafit Plus cementless liner and the Biolox delta acetabular cup all by B Braun Medical Ltd. The participating consultant routinely uses computer aided orthopaedic surgery (CAOS) techniques to implant the stem and the acetabular cup and all study patients will have surgery using these techniques.

Participants will have their standard in-patient care and rehabilitation. Standard hospital practice for hip arthroplasty patients is for them to return to the hospital for a post-operative review at three months. During this appointment they will be reviewed by a member of the arthroplasty team and have two radiographs taken, an anterior/posterior view of the full pelvis and a lateral view of the index hip. Study participants will return for the three month post-operative review and be seen by the arthroplasty team as standard, but will not have the two radiographs taken. Instead, they will have a computed tomography (CT) scan taken of the full pelvis. In addition to the standard clinical outcome data collected, Participants will also complete the Harris Hip Score and a range of motion questionnaire. Study participants will also have an additional assessment as part of their three month post-operative review. In the movement analysis laboratory in the Golden Jubilee National Hospital, they will undergo a RoM assessment using clinical movement analysis techniques. During this assessment, participants will be asked to fully flex/extend their hip joint, fully abduct/adduct it, fully internally/externally rotate it and finally fully circumduct it. While performing these tasks, their hip joint movement will be tracked by a number of infrared cameras identifying small reflective markers attached to their body. A computer can convert these data into three dimensional RoM data for further analysis. At the end of their three month post-operative review, the participant's involvement in the study will be complete.

The computer used for CAOS is capable of measuring the on-table range of motion (RoM) of the hip. This data will be collected for the purposes of the study. Mathematical methods will be used to determine the theoretical RoM of the hip from the CT scan. The data from the movement analysis session will give the actual RoM. The CT scan will be analysed to determine the inclination and version of the acetabular cup and the torsion of the femoral stem. From this, the combined anteversion (CA) of the cup/stem system will be determined. Comparison will be made between the CA and the actual RoM to determine to what extent, if any, the CA influences the RoM. Comparisons will be made between the on-table RoM and the theoretical RoM, and the actual RoM to assess the accuracy of the methods used to determine the on-table and theoretical RoMs.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty under the care of the participating consultant
* Males and females aged between 55 and 80 years
* Willing to return for the follow-up appointment
* Willing to take part
* Able to give informed consent

Exclusion Criteria:

* Revision total hip arthroplasty
* Second stage of staged bilateral total hip arthroplasty if already recruited for the first stage
* Males over 70 years (as per participating surgeon's standard practice for the Excia T stem)
* Females who are pregnant
* Not suitable to receive an Excia T stem, a Plasmacup or a ceramic head

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Actual hip range of movement in degrees measured using clinical movement analysis | Three months
  Hip RoM in three dimensions measured using clinical movement analysis techniques

SECONDARY OUTCOMES:
Theoretical hip range of movement in degrees calculated from CT scans | Three months
  Hip RoM in three dimensions determined mathematically from the CT scan
On-table hip range of movement in degrees as measured by the operative navigation computer | Intra-operatively
  Hip RoM in three dimensions measured using the CAOS computer system
Combined anteversion in degrees of the acetabular cup and femoral stem system measured from CT scans | Three months
  A measure of the hip implant orientation using the torsion of the stem and the version of the cup
Leg length discrepancy | Three months
  difference in leg length measured from the CT scan
Oxford Hip Score | Three months
  Patient reported hip pain and function
EQ-5D | Three months
  Patient reported quality of life
Harris Hip Score | Three months
  Clinician assessed hip pain and function
Patient satisfaction measured on a five point Likert scale | Three months
  Patient reported satisfaction with hip
Number of dislocations in cohort | Three months
  Post-operative dislocations
Number of revisions in cohort | Three months
  Revision rate
Number of infections in cohort | Three months
  Post-operative surgical site infections
Operative time in minutes | Intra-operative
  Length of operation
Blood loss volume | Intra-operative
  Amount of blood lost
Blood transfusion (Yes/No) | Intra-operative
  Peri-operative blood transfusion data

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Deep, M.D., Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No